CLINICAL TRIAL: NCT04348656
Title: A Randomized Open-Label Trial of CONvalenscent Plasma for Hospitalized Adults With Acute COVID-19 Respiratory Illness (CONCOR-1)
Brief Title: CONvalescent Plasma for Hospitalized Adults With COVID-19 Respiratory Illness (CONCOR-1)
Acronym: CONCOR-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated after the planned interim analysis as the pre-defined futility threshold was met
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Blood Services (Other); Héma-Québec (Other); University of Toronto (Other); Université de Montréal (Other); Weill Medical College of Cornell University (Other); New York Blood Center (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONCOR-1; NCT04418518 (obsolete NCT alias)
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Convalescent plasma; Transfusion; SARS-CoV-2; Passive immunization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convalescent plasma (Experimental): ~500 mL ABO compatible convalescent apheresis plasma
  Interventions: Biological: Convalescent plasma
- Standard of care (No Intervention): Treated as per institutional standard of care.

INTERVENTIONS:
Biological: Convalescent plasma — Patients will receive 500 mL of convalescent plasma (from one single-donor unit of 500 mL or 2 units of 250 mL from 1-2 donations) collected by apheresis from donors who have recovered from COVID-19 and frozen (1 year expiration date from date of collection). The plasma unit will be thawed as per standard blood bank procedures and infused into the patient slowly over 4 hours. When administering 2 units of 250 mL, the 2nd unit will be administered after the first, and no longer than 12 hours later. The patient will be monitored for adverse events as per each site's policies.
  Arms: Convalescent plasma

SUMMARY:
There is currently no treatment available for COVID-19, the acute respiratory illness caused by the novel SAR-CoV-2. Convalescent plasma from patients who have recovered from COVID-19 that contains antibodies to the virus is a potential therapy. On March 25th, 2020, the FDA approved the use of convalescent plasma under the emergency investigational new drug (eIND) category. Randomized trials are needed to determine the efficacy and safety of COVID-19 convalescent plasma for acute COVID-19 infection.

The objective of the CONCOR-1 trial is to determine the efficacy of transfusion of COVID-19 convalescent plasma to adult patients admitted to hospital with COVID-19 infection at decreasing the frequency of in-hospital mortality in patients hospitalized for COVID-19.

It is hypothesized that treating hospitalized COVID-19 patients with convalescent plasma early in their clinical course will reduce the risk of death, and that other outcomes will be improved including risk of intubation, and length of ICU and hospital stay.

This pan-Canadian clinical trial has the potential to improve patient outcomes and reduce the burden on health care resources including reducing the need for ICU beds and ventilators.

DETAILED DESCRIPTION:
Problem to be addressed: In December 2019, the Wuhan Municipal Health Committee (Wuhan, China) identified an outbreak of viral pneumonia cases of unknown cause. Coronavirus RNA was quickly identified in some of these patients.This novel coronavirus has been designated SARS-CoV-2, and the disease caused by this virus has been designated COVID-19.Outbreak forecasting and mathematical modelling suggest that these numbers will continue to rise [1] in many countries over the coming weeks to months.Global efforts to evaluate novel antivirals and therapeutic strategies to treat COVID-19 have intensified. There is an urgent public health need for rapid development of novel interventions. At present, there is no specific antiviral therapy for coronavirus infections.

Passive immunization:Passive immunization consists in the transfer of antibodies from immunized donor to non-immunized individual in order to transfer transient protection against an infective agent. A physiological example of passive immunization is the transfer of maternal IgG antibodies to the foetus through the placenta to confer humoral protection to newborns in the first years of life. Passive immunization differs from active immunization in which the patient develops their own immune response following contact with the infective agent or vaccine.

Known potential risks and benefits: There is a theoretical risk of antibody-dependent enhancement of infection (ADE) through which virus targeted by non-neutralizing antibodies gain entry into macrophages. Another theoretical risk is that antibody administration to those exposed to SARS-CoV-2 may avoid disease but modify the immune response such that those individuals mount attenuated immune responses, which would leave them vulnerable to subsequent re-infection. Finally, there are risks associated with any transfusion of plasma including transmission of blood transmitted viruses (e.g. HIV, HBV, HCV, etc.), allergic transfusion reactions, including anaphylaxis, febrile non hemolytic transfusion reaction, transfusion related acute lung injury (TRALI), transfusion associated cardiac overload (TACO), and hemolysis should ABO incompatible plasma be administered. Potential benefits of COVID-19 convalescent plasma include improved survival, improvement in symptoms, decreased risk in intubation for mechanical ventilation, decrease risk of intensive care unit (ICU) admission, shortened hospitalization time and suppression of viral load.

Mechanism of action: Transfusion of apheresis frozen plasma (AFP) from COVID-19 convalescent patients allows the transfer of donor neutralizing antibodies directed against SARS-CoV2 antigens to the recipient, thus allowing the generation of passive immunization. Naturally produced human antibody are polyclonal, meaning they are directed against a variety of different viral antigens and epitopes allowing for a general neutralizing effect against the virus rather than focussing on a specific target. Administration of convalescent plasma has been associated with rapid decrease in viral load. It is also possible that passive immunization contributes to improved cell-mediated immunity by favoring the phagocytosis and presentation of viral antigens to host T cells.

Participant recruitment:Only hospitalized COVID-19 patients are eligible so recruitment efforts will be focused on identified consecutive patients admitted to hospital with acute COVID-19 infection. No other external recruitment efforts are planned. At each participating hospital, a process for identifying patients with COVID-19 will be established.

Donor recruitment for Canadian sites: Recovered COVID-19 patients will be identified as potential donors in collaboration with provincial public health services, local health authorities, and individual co-investigators involved in the study. Potential donors may also be recruiting following self-identification on the routine donor questionnaire or through social media. They will be contacted by phone and invited to participate in the program as potential donors. After obtaining verbal consent and reviewing donor selection criteria, eligible participants will be directed to a Héma-Québec collection or Canadian Blood Services apheresis collection site in their area to donate.

Criteria for donors: All donors will need to meet the criteria set forth in the Manual of donor selection criteria in use at Héma-Québec or Canadian Blood ServicesIn addition, donors will require:

* Prior diagnosis of COVID-19 documented by a PCR test at time of infection or by positive anti-SARS-CoV-2 serology following infection
* Male donors, or female donors with no pregnancy history or with negative anti-HLA antibodies
* At least 6 days since last plasma donation
* Provided informed consent
* A complete resolution of symptoms at least 14 days prior to donation

Donor recruitment for United States sites: Recovered COVID-19 patients are being recruited through the New York Blood Center and Weill Cornell Medicine in separate protocols. Potential donors can self-refer via websites but also be referred by physicians or identified via the medical record system. Only donors with laboratory-confirmed history of COVID-19 will be screened. After providing consent and reviewing FDA and NYBC donor eligibility criteria, donors are screened for the presences of SARS-CoV-2 virus in the nasopharynx if screening within 14 days of complete resolution in accordance with current FDA guidance. Criteria for donation are subject to change based on future revision of FDA guidance. Those found to be eligible will be referred to NYBC for donation.

Criteria for donors:

* Provision of informed consent
* Aged 18 to 70 years. Donors are not longer eligible after their 71st birthday.
* Documented molecular diagnosis of SARS-CoV-2 by RT-PCR by nasopharyngeal swab, oropharyngeal swab, or sputum or detection of anti-SARS-CoV-2 IgG in serum.
* Complete resolution of COVID-19 symptoms at least 14 days prior to donation
* Not currently pregnant or pregnant within 6 weeks by self-report
* Male donors, or females with no pregnancy history or with negative anti-HLA antibodies
* Meets blood donor criteria specified by NYBC, which is consistent with FDA regulations.

Donors will be allowed to donate every 7 days. The following information will be collection from donors: ABO group, sex, age, date of onset of symptoms (when available), date of resolution of symptoms (when available), CCP collection date(s).

Randomization procedures: Patients will be randomized in a 2:1 ratio (convalescent plasma vs standard of care). Patients will be randomized using a secure, concealed, computer-generated, web-accessed randomization sequence. Randomization will be stratified by centre and age (<60 and ≥ 60 years). Within each stratum, variable permuted block sized will be used. This approach will ensure that concealment of the treatment sequence is maintained.

Duration of follow-up: Subjects will be followed daily until hospital discharge or death. Patients discharged from hospital before Day 30 will be contacted by telephone on Day 30 ± 3 days to ascertain any AEs, vital status (dead/alive), hospital readmission and need for mechanical ventilation after discharge. Patients discharged from hospital will be contacted at Day 90+/- 7 days to determine vital status. Patients with a prolonged hospital admission will be censored at Day 90. The local study coordinator will collect all study data and record the data in the electronic CRF or paper CRF as per study procedures for each site.

Duration of study: For an individual subject, the study ends 90 days after randomization. The overall study will end when the last randomized subject has completed 90 day follow-up. We estimate that all patient will be enrolled in a period of 6 months, data on the primary endpoint will be available 30 days after last patient enrollment and data on all secondary endpoints will be available after 90-day from last patient enrollment.

Sample size considerations: Assuming a baseline risk of intubation or death of 30% in hospitalized patients with standard of care, a sample size of 1200 (800 in the convalescent plasma arm, and 400 in the standard of care arm) would provide 80% power to detect a relative risk reduction of 25% with convalescent plasma therapy using a 2-tailed test at level α = 0.05 and a 2:1 randomization.

Interim analysis: A single interim analysis is planned when the primary outcome (intubation or mortality at 30 days) is available for 50% of the target sample. An O'Brien-Fleming stopping rule will be used at that time, but treated as a guideline, so there is minimal impact on the threshold for statistical significance for the final significance test of the primary outcome. A DSMB will monitor ongoing results to ensure patient well-being and safety as well as study integrity. The DSMB will be asked to recommend early termination or modification only when there is clear and substantial evidence of a treatment difference.

Final analysis plan: The primary analysis will be based on the intention-to-treat population which will include data from all individuals who have been randomized. Outcomes will be attributed to the arm to which individuals were randomized irrespective of whether they received the planned intervention (e.g. plasma from a convalescent COVID-19 donor).

ELIGIBILITY:
Inclusion Criteria:

* ≥16 years old (>18 years of age in the United States)
* Admitted to hospital with confirmed COVID-19 respiratory illness
* Receiving supplemental oxygen
* 500 mL of ABO compatible convalescent plasma is available

Exclusion Criteria:

* Onset of respiratory symptoms >12 days prior to randomization
* Intubated or plan in place for intubation
* Plasma is contraindicated (e.g. history of anaphylaxis from transfusion)
* Decision in place for no active treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2020-03-14 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Arnold, MD, Principal Investigator — McMaster University
Locations (73):
- United States (3):
  - Brooklyn Hospital, Brooklyn, New York
  - Lower Manhattan Hospital, New York, New York
  - Weill Cornell Medical Center, New York, New York
- Brazil (2):
  - Hospital Universitário Antônio Pedro (HUAP), Niterói
  - Hemario, Rio de Janeiro
- Canada (68):
  - Peter Lougheed Center, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - University of Alberta - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta
  - Fraser Health Authority - Abbotsford Regional Hospital and Cancer Centre, Abbotsford, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Grace General Hospital, Winnipeg, Manitoba
  - Vitalité Health Network - Acadie-Bathurst, Bathurst, New Brunswick
  - Vitalité Health Network - Restigouche, Campbellton, New Brunswick
  - Vitalité Health Network- Northwest, Edmundston, New Brunswick
  - Dr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick
  - Lakeridge Health Ajax Pickering, Ajax, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - St. Mary's Hospital, Kitchener, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Partners - Mississauga Hospital, Mississauga, Ontario
  - Trillium Health Partners - Credit Valley, Mississauga, Ontario
  - North York General Hospital, North York, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Queensway Carleton Hospital, Ottawa, Ontario
  - Niagara Health System - St. Catherines, Saint Catherines, Ontario
  - Bluewater Health, Sarnia, Ontario
  - Scarborough Health Network, Centenary Hospital, Scarborough Village, Ontario
  - Scarborough Health Network, General Hospital, Scarborough Village, Ontario
  - Scarborough Health Network, Birchmount Hospital, Scarborough Village, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health St. Michael's Hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Unity Health, St. Joseph's Health Care Centre, Toronto, Ontario
  - Windsor Regional Hospital - Metropolitan Campus, Windsor, Ontario
  - Windsor Regional Hospital - Ouellette Campus, Windsor, Ontario
  - L'Hopital Chicoutimi, Chicoutimi, Quebec
  - Hôpital de la Cité-de-la-Santé, Laval, Quebec
  - Hotel Dieu Hospital of Lévis, Lévis, Quebec
  - Hôpital Charles-Le Moyne, Longueuil, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Montréal General Hospital, Montreal, Quebec
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire (CHU) de Québec - Université Laval, Québec, Quebec
  - Institut Universitaire de cardiologie et pneumologie de Québec, Québec, Quebec
  - Centre hospitalier régional de St-Jérôme, Saint-Jérôme, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS) - Hôpital Hôtel-Dieu, Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS) - Hôpital Fleurimont, Sherbrooke, Quebec
  - Centre hospitalier affilié universitaire régional de Trois-Rivières, Trois-Rivières, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Pasqua Hospital, Regina, Saskatchewan
  - St. Paul's Hospital, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JT, Leung K, Leung GM. Nowcasting and forecasting the potential domestic and international spread of the 2019-nCoV outbreak originating in Wuhan, China: a modelling study. Lancet. 2020 Feb 29;395(10225):689-697. doi: 10.1016/S0140-6736(20)30260-9. Epub 2020 Jan 31. PMID 32014114
- [Background] 2. FDA USFDA. Investigational COVID-19 Convalescent Plasma - Emergency INDs [Web]. 2020 [Available from: https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-device-exemption-ide-process-cber/investigational-covid-19-convalescent-plasma-emergency-inds accessed March 26th 2020.
- [Derived] Begin P, Callum J, Jamula E, Cook R, Heddle NM, Tinmouth A, Zeller MP, Beaudoin-Bussieres G, Amorim L, Bazin R, Loftsgard KC, Carl R, Chasse M, Cushing MM, Daneman N, Devine DV, Dumaresq J, Fergusson DA, Gabe C, Glesby MJ, Li N, Liu Y, McGeer A, Robitaille N, Sachais BS, Scales DC, Schwartz L, Shehata N, Turgeon AF, Wood H, Zarychanski R, Finzi A; CONCOR-1 Study Group; Arnold DM. Convalescent plasma for hospitalized patients with COVID-19: an open-label, randomized controlled trial. Nat Med. 2021 Nov;27(11):2012-2024. doi: 10.1038/s41591-021-01488-2. Epub 2021 Sep 9. PMID 34504336
- [Derived] Begin P, Callum J, Heddle NM, Cook R, Zeller MP, Tinmouth A, Fergusson DA, Cushing MM, Glesby MJ, Chasse M, Devine DV, Robitalle N, Bazin R, Shehata N, Finzi A, McGeer A, Scales DC, Schwartz L, Turgeon AF, Zarychanski R, Daneman N, Carl R, Amorim L, Gabe C, Ellis M, Sachais BS, Loftsgard KC, Jamula E, Carruthers J, Duncan J, Lucier K, Li N, Liu Y, Armali C, Kron A, Modi D, Auclair MC, Cerro S, Avram M, Arnold DM. Convalescent plasma for adults with acute COVID-19 respiratory illness (CONCOR-1): study protocol for an international, multicentre, randomized, open-label trial. Trials. 2021 May 4;22(1):323. doi: 10.1186/s13063-021-05235-3. PMID 33947446
- See also: Publication of trial results in Nature Medicine — https://www.nature.com/articles/s41591-021-01488-2

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Plasma | Standard of Care
Started | 627 | 313
Baseline Population | 625 | 313
Intention to Treat Analysis | 614 | 307
Per Protocol Analysis | 548 | 303
Completed | 614 | 307
Not Completed | 13 | 6
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Plasma | Standard of Care | Total
Number analyzed (Participants) | 625 | 313 | 938
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (16.0) | 67.1 (14.8) | 67.5 (15.6)
Age, Customized [Count of Participants; unit: Participants]
  >= 60 years | 438 | 218 | 656
  < 60 years | 187 | 95 | 282
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 256 | 128 | 384
  Male | 369 | 185 | 554
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 305 | 153 | 458
  Asian | 104 | 46 | 150
  Hispanic or Latino | 34 | 9 | 43
  Black | 25 | 11 | 36
  Other | 38 | 28 | 66
  Unknown | 119 | 66 | 185
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 529 | 265 | 794
  United States | 89 | 45 | 134
  Brazil | 7 | 3 | 10
Pregnancy present at randomization [Count of Participants; unit: Participants] | 4 | 1 | 5
ABO blood group [Count of Participants; unit: Participants]
  O | 270 | 113 | 383
  A | 235 | 121 | 356
  B | 89 | 57 | 146
  AB | 31 | 22 | 53
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: 259 patients (171 in the convalescent plasma arm and 88 in the standard of care arm) had an unknown BMI and were not included in this analysis.
  kg/m^2
    number analyzed (Participants) | 454 | 225 | 679
    (all) | 30.0 (7.5) | 30.0 (7.4) | 30.0 (7.4)
Body Mass Index [Count of Participants; unit: Participants]
  BMI < 30 kg/m^2 | 256 | 123 | 379
  BMI >= 30 kg/m^2 | 198 | 102 | 300
  BMI Unknown | 171 | 88 | 259
Presence of comorbidity [Count of Participants; unit: Participants]
  Diabetes | 220 | 108 | 328
  Cardiac disease | 385 | 197 | 582
  Baseline respiratory diseases | 147 | 79 | 226
Abnormal CT chest or chest x-ray result before randomization [Count of Participants; unit: Participants] | 563 | 266 | 829
Medication for other research study at baseline [Count of Participants; unit: Participants] | 53 | 41 | 94
Medication for COVID-19 at baseline [Count of Participants; unit: Participants]
  Azithromycin | 279 | 137 | 416
  Other antibiotics | 405 | 186 | 591
  Systemic corticosteroids | 496 | 258 | 754
  Antiviral medications | 165 | 80 | 245
  Anticoagulants | 355 | 180 | 535
  Other COVID-19 medications | 79 | 39 | 118
Medication not for COVID-19 at baseline [Count of Participants; unit: Participants]
  Angiotensin-converting enzyme inhibitor | 85 | 63 | 148
  Angiotensin-converting enzyme receptor blocker | 77 | 47 | 124
  Non-steroidal anti-inflammatory drugs | 77 | 52 | 129
  Colchicine | 5 | 2 | 7
  Systemic corticosteroids | 61 | 35 | 96
  Inhaled corticosteroids | 84 | 42 | 126
  Immunomodulatory agents | 22 | 18 | 40
  Anticoagulants | 135 | 64 | 199
Systemic corticosteroid at baseline [Count of Participants; unit: Participants] | 504 | 262 | 766
Fraction of inhaled oxygen (FiO2) at the time of randomization [Mean (Standard Deviation); unit: percentage of oxygen] — FiO2 is an estimation of the oxygen content (% of oxygen) in the air that a person inhales. Use of supplemental oxygen (eg. through nasal prongs, an oxygen mask, intubation, etc) increases the oxygen content of the inhaled air.
  percentage of oxygen | 49.5 (25.2) | 48.8 (25.1) | 49.3 (25.2)
Time from any symptom onset to randomization [Mean (Standard Deviation); unit: days] | 8.0 (3.8) | 7.8 (3.4) | 7.9 (3.7)
Time from COVID-19 diagnosis to randomization [Mean (Standard Deviation); unit: days] — COVID-19 diagnosis is defined as the date of positive COVID-19 test
  days | 4.9 (3.6) | 5.1 (4.4) | 5.0 (3.9)
Location at time of randomization [Count of Participants; unit: Participants]
  Ward | 505 | 260 | 765
  Intensive care unit | 120 | 53 | 173
Enrolled in other clinical trials [Count of Participants; unit: Participants] | 168 | 98 | 266

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Intubated or Died
Description: Endpoint of the need for intubation or patient death
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
Participants | 199 | 86
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.18, wald test; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.94 to 1.43]

2. Secondary Outcome: Time to Intubation or In-hospital Death
Description: Time in days from randomization to occurrence of intubation or death
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
days | 22.8 (11.0) | 23.4 (11.0)
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.30, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.89 to 1.47]

3. Secondary Outcome: Ventilator-free Days by Day 30
Description: Number of days off ventilator at 30 days
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
days | 23.4 (10.4) | 24.0 (10.5)
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.41, t-test, 2 sided; bootstrap estimates based on resampling process; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.1 to 0.7] — bootstrap estimates based on resampling process

4. Secondary Outcome: Death by Day 30
Description: Occurrence of patient death at 30 days
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
Participants | 141 | 63
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.40, wald test; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.86 to 1.46]

5. Secondary Outcome: Length of Stay in Intensive Care Unit (ICU)
Description: Number of days spent in the intensive care unit (ICU) over the 30-day period following randomization
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
days | 4.3 (7.9) | 3.7 (7.1)
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.3 to 1.7]

6. Secondary Outcome: Need for Renal Replacement Therapy
Description: Need for new renal replacement therapy
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available. Data from 11 patients on chronic kidney replacement therapy at baseline were not included in the Count of Participants since they were receiving renal replacement therapy prior to study entry and therefore do not meet our criteria for needing new renal replacement therapy during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
Participants | 10 | 6
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.72, t-test, 2 sided; bootstrap estimates based on resampling process; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.31 to 2.27] — bootstrap estimates based on resampling process

7. Secondary Outcome: Need for Extracorporeal Membrane Oxygenation (ECMO)
Description: Requirement for extracorporeal membrane oxygenation (ECMO)
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
Participants | 0 | 1

8. Secondary Outcome: Development of Myocarditis
Description: New diagnosis of myocarditis
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
Participants | 0 | 0

9. Secondary Outcome: In-hospital Death
Description: Occurrence of death while in hospital, censored at 90 days. Patients who were still in hospital at Day 30 were followed until Day 90 to capture in-hospital mortality.
Time Frame: Day 90
Population: Baseline study population- all randomized patients, excluding 2 who withdrew consent prior to the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 625 | 313
Participants | 156 | 69
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.33, wald test; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.88 to 1.45]

10. Secondary Outcome: Time to In-hospital Death
Description: Time to in-hospital death at 90 days. Patients who were still in hospital at Day 30 were followed until Day 90 to capture in-hospital mortality.
Time Frame: Day 90
Population: Baseline study population (all randomized patients, excluding 2 who withdrew consent prior to the intervention)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 625 | 313
days | 16.3 (17.1) | 14.8 (16.3)
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.91, Regression, Cox; competing risk analysis; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.76 to 1.35] — competing risk analysis

11. Secondary Outcome: Length of Stay in Hospital
Description: Number of days from randomization to death or hospital discharge. Patients still in hospital at Day 30 were followed until Day 90 to capture death or discharge from hospital.
Time Frame: Day 90
Population: Baseline study population- all randomized patients, excluding 2 who withdrew consent prior to receiving the intervention
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 625 | 313
days | 16.3 (17.1) | 14.8 (16.3)
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.18, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.80 to 1.04]

12. Secondary Outcome: Number of Participants With Grade 3 and 4 Serious Adverse Events
Description: Number of participants with Grade 3 and 4 (CTCAE v4.0) serious adverse events, and cumulative incidence of Grade 3 and 4 serious adverse events (using MedDRA AE terms)
Time Frame: Day 30
Population: Intention to treat population with data on the primary outcome available
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
Participants | 92 | 30
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.03, wald test; Risk Ratio (RR) = 1.53, 95% CI 2-sided [1.04 to 2.26]
Statistical Analysis 2: Comparison: Convalescent Plasma vs Standard of Care; The cumulative incidence of Grade 3 and 4 serious AEs is described as a hazard ratio; Test type: Superiority; p = 0.02, Regression, Cox; competing risk analysis; Hazard Ratio (HR) = 1.70, 95% CI 2-sided [1.08 to 2.69] — competing risk analysis

13. Secondary Outcome: Number of Participants With CCP Transfusion-associated Adverse Events (AE)
Description: Number of participants experiencing CCP transfusion-associated adverse events (AE), as defined by the International Society of Blood Tranfusion (ISBT ) classification
Time Frame: Day 30
Population: Only patients in the convalescent plasma (CCP) arm (intention to treat population) are assessed for CCP-related transfusion events, as these cannot occur in the standard of care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 0
Participants | 35 | 0

14. Secondary Outcome: Number of Participants With Grade 3, 4, or 5 Serious Adverse Events
Description: Number of Participants with Grade 3-5 (CTCAE v4.0) serious adverse events reported to Day 30
Time Frame: Day 30
Population: Intention to treat population with data on primary outcome available
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 614 | 307
Participants | 205 | 81
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Superiority; p = 0.03, wald test; Risk Ratio (RR) = 1.27, 95% CI 2-sided [1.02 to 1.57]

15. Secondary Outcome: Patient Reported Outcome Using Change in EQ-5D-5L Score
Description: Change in score on EQ-5D-5L instrument at Day 30 as compared to baseline. The EQ-5D-5L measures health-related quality of life in five dimensions, namely, mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients can report five level impairment, reflecting no, slight, moderate, severe, and extreme problems in each dimension. The range of possible values is -0.148 to 0.949, with a higher score reflecting a better outcome. For the change in score, a positive number indicates that the scores improved from baseline.
Time Frame: Baseline and Day 30
Population: Patients with a complete EQ-5D-5L at both baseline AND Day 30. Patients who were unable to complete the EQ-5D-5L due to their health status or other reason are excluded from this population. Proper administration of the EQ-5D-5L requires the answers be obtained directly from the patient.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 272 | 157
units on a scale | 0.150 (0.2588) | 0.157 (0.2859)

16. Secondary Outcome: Patient Reported Outcome- Quality-adjusted Life Days
Description: Quality-adjusted life days calculated using the EQ-5D-5L score. Quality-adjusted life days is a measure of how well a patient lives for how long. It combines the length of life and quality of life into one value. This is calculated by multiplying the health utility (derived from the EQ-5D-5L score) by the amount of time the patient is alive during the study period. A higher number is better.
Time Frame: Day 30
Population: Patients with a completed baseline EQ-5D-5L AND either a completed EQ-5D-5L at Day 30 or who were dead at Day 30. Patients who did not have a completed baseline EQ-5D-5L were excluded from this population.
Measure: Mean (Standard Deviation); unit: quality adjusted life days
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 341 | 194
quality adjusted life days | 17.959 (9.0363) | 18.037 (8.9771)

17. Secondary Outcome: Cost of Intervention and Hospital Stay
Description: Cost per patient calculated using cost of the intervention and costs of the hospital stay
Time Frame: Day 30
Population: Patients with a completed baseline EQ-5D-5L AND either a completed EQ-5D-5L at Day 30 or who were dead at Day 30. The cost results will be combined with the quality-adjusted life day results to calculate the incremental cost per quality-adjusted life day, so the analysis population matches that of the quality-adjusted life day analysis.
Measure: Mean (Standard Deviation); unit: Canadian dollars
Arm/Group | Convalescent Plasma | Standard of Care
Number analyzed (Participants) | 341 | 194
Canadian dollars | 23516.74 (21373.80) | 20025.05 (17957.57)
Statistical Analysis 1: Comparison: Convalescent Plasma vs Standard of Care; Test type: Other — Incremental cost per quality-adjusted life day gained (ICER)- this is a summary measure of the cost-effectiveness of the intervention, compared to the control group. This is calculated using the cost (derived from cost of the intervention and cost of hospital stay based on the payer's perspective) per patient and the quality-adjusted life days calculated using the EQ-5D-5L results; ICER (CAD) = -44623.01, 95% CI 2-sided [-525369.24 to 436123.22] — ICER is reported in Canadian dollars. 95% CI is calculated by 1000 bootstrap sampling using bias-corrected accelerated method

ADVERSE EVENTS:
Time Frame: AEs: 30 days; any death (in-hospital or otherwise): 30 days. Participants still in hospital at 30 days were followed for 90 days for in-hospital death only (no AE collection and no follow up once discharged past Day 30).
Description: MedDRA 12.1 was used for AE terminology jointly with CTCAE v4.0 for AE severity grading.
  Serious and Other (Not Including Serious) Adverse Events assessed for the Intention to Treat Population and All-Cause Mortality assessed for the Baseline Population.
  The number of deaths reported under "all cause mortality" include all reported deaths prior to Day 30, plus any in-hospital deaths occurring up to Day 90 in patients who were still in hospital at Day 30.
Arm/Group | Convalescent Plasma | Standard of Care
All-Cause Mortality (participants affected / at risk) | 160/625 | 70/313
Serious Adverse Events (participants affected / at risk) | 205/614 | 81/307
Other Adverse Events (participants affected / at risk) | 110/614 | 35/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Plasma (N=614) | Standard of Care (N=307)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 70 | 33
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 57 | 22
Acute kidney injury (Renal and urinary disorders) | 12 | 7
Death NOS (General disorders) | 14 | 4
Sepsis (Infections and infestations) | 11 | 5
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Lung infection (Infections and infestations) | 6 | 4
Multi-organ failure (General disorders) | 6 | 3
Hypotension (Vascular disorders) | 8 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Thromboembolic event (Vascular disorders) | 4 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Cardiac arrest (Cardiac disorders) | 3 | 2
Asystole (Cardiac disorders) | 4 | 0
Infections and infestations - Other (Infections and infestations) | 3 | 1
Intracranial hemorrhage (Nervous system disorders) | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Transfusion associated circulatory overload (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — TACO is characterized by any four of the following: acute respiratory distress, tachycardia, increased blood pressure, acute or worsening pulmonary edema on chest xray, evidence of positive fluid balance within 6h of completion of transfusion
Anemia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Delirium (Psychiatric disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 0
Stroke (Nervous system disorders) | 0 | 2
Transfusion associated dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Respiratory distress within 24h of transfusion that does meet criteria for TACO, TRALI, or allergic reaction. Respiratory distress should be the most prominent clinical feature and should not be explained by the pt's condition or another known cause
Possible transfusion related acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — In patients with no acute lung injury prior to transfusion, a new acute lung injury meeting ISBT criteria that is present during or within 6 hours of transfusion.
Cardiac disorders - Other (Cardiac disorders) | 1 | 0
Cardiac troponin T increased (Investigations) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
CPK increased (Investigations) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Pregnancy, puerperium and perinatal conditions - Other (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urine output decreased (Renal and urinary disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Plasma (N=614) | Standard of Care (N=307)
Lymphocyte count decreased (Investigations) | 17 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 18 | 6
Infections and infestations, other (Infections and infestations) | 13 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 5
Anemia (Blood and lymphatic system disorders) | 14 | 3
Hypertension (Vascular disorders) | 11 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 9 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 8 | 1
Urinary tract infection (Infections and infestations) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04348656/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT04348656/SAP_001.pdf